CLINICAL TRIAL: NCT06278207
Title: Finerenone Research of Outcomes and Drug Utilization
Brief Title: An Observational Study Called FINEROD to Learn More About the Use of the Treatment Finerenone Including How Safe it is and How Well it Works Under Real-world Conditions
Acronym: FINEROD
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22731
Record Dates: First submitted 2024-02-09; First posted 2024-02-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with CKD and T2D who initiate finerenone: The data sources used include a network of commercial electronic health records (EHRs) and national claims data in Asia and in the United States.
  Interventions: Drug: Finerenone (BAY 94-8862)

INTERVENTIONS:
Drug: Finerenone (BAY 94-8862) — 10 mg or 20 mg daily
  Other Names: Kerendia, Firialta

SUMMARY:
This is an observational study, in which data from people in Asia and in the United States with chronic kidney disease (CKD) together with type 2 diabetes (T2D) are studied. The participants in this study are already receiving the study treatment finerenone as part of their regular care from their doctors. In observational studies, only observations are made without specified advice or interventions. CKD is a long-term progressive decrease in the kidneys' ability to work properly. In people with T2D, the body does not make enough of a hormone called insulin, or does not use insulin well enough. The resulting high blood sugar levels can cause damage to the kidneys. CKD often occurs together with T2D or as a consequence of T2D. Finerenone works by blocking certain proteins, called mineralocorticoid receptors. By doing this, it may reduce damage to kidneys, heart and blood vessels. Finerenone was recently approved in the US and is now available for doctors to prescribe to people with CKD together with T2D. Consequently, there is a need to collect more information about how finerenone is used, its safety and how well it works under real-world conditions. The main purpose of this study is to collect and describe the characteristics of people with CKD and T2D who are receiving initiate finerenone treatment as prescribed by their doctors. To do this, the researchers will collect general information of the participants such as age or gender and data on kidney function and possible heart problems.

The researchers will also collect data on any other disease or medical condition in the participants and on other medications used while taking finerenone.

The data will come from a network of commercial electronic health records (EHRs) and national claims data in the United States and in Asia. They cover the period from July 1st, 2021 until the latest data cut available for each dataset. Only already available data is collected and studied. There are no required visits or tests in this study.

ELIGIBILITY:
Inclusion Criteria:

* A minimum of 12 months of continuous enrolment in the databases with medical and pharmacy coverage measured as continuously receiving medical care from health providers contributing to the EHR or claims system, depending on the database used
* No recorded prescription for finerenone in the 12 months prior to the index date
* Age of 18 years or older as of the index date
* Evidence of T2D at any point before (and including) the index date.
* CKD stages 2-4 related to eligibility will be defined according to the presence of the following criteria at any point before (and including) the index date:

  * A diagnosis code indicating CKD stage 2, 3, 4 or stage unspecified
  * two UACR tests results ≥ 30 mg/g separated by at least 90 days and by not more than 540 days
  * two different eGFR test results ≥ 15 mL/min/1.73 m2 AND < 60 mL/min/1.73 m2 separated by at least 90 days and by not more than 540 days

Exclusion Criteria:

- Kidney failure defined as follows:

* Two different eGFR test results < 15 mL/min/1.73 m2 separated by at least 90 days and by not more than 540 days;
* Dependence on dialysis (at least 3 sessions over at least 90 days during the baseline period);
* A diagnosis code indicating kidney failure or CKD stage 5; Kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic kidney disease and type 2 diabetes who initiate finerenone in secondary data sources (electronic health records (EHR) and claims data) in the United States and in Asia.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Participants' characteristics at baseline in a cohort of participants with CKD and T2D who initiate finerenone. | 12 months before first prescription/dispensation of finerenone (index date)
  Sociodemographic characteristics such as age, sex, race and socio-economic status.
Participants' comorbidities at baseline in a cohort of participants with CKD and T2D who initiate finerenone. | 12 months before first prescription/dispensation of finerenone (index date)
  Including heart diseases, lipid diseases, liver disease, hospitalization for acute kidney injury, dementia, body mass index, smoking status, alcohol abuse, and other comorbidities measured using comorbidities indexes (such as the Charlson comorbidity index)
Participants' comedications at baseline in a cohort of participants with CKD and T2D who initiate finerenone. | 12 months before first prescription/dispensation of finerenone (index date)
  In subcohorts of participants in co-medication between finerenone and other hypertensive and diabetic medications (SGLT2i, RAASi, GLP-1 RA, etc.), characterized by CKD stage, including a 15-25 ml/min/1.73 m2 eGFR subgroup.

SECONDARY OUTCOMES:
Proportion of finerenone initiators with and without UACR measurements at baseline | From first prescription/dispensation of finerenone (index date) until 12 months after index date
  UACR=Urinary Albumin-to-Creatinine Ratio
Average UACR in the subcohort with UACR measurements | From first prescription/dispensation of finerenone (index date) until 12 months after index date
Incidence rate of kidney failure in participants with CKD and T2D that initiate finerenone. | From first prescription/dispensation of finerenone (index date) until end of follow-up (death, disenrollment, development of either kidney failure or kidney cancer, or by the last available date in the corresponding database) up to 150 months
  Any of the following:
  ≥ 2 outpatient eGFR measurements of < 15 mL/min/1.73 m2 separated by at least 90 days; Record of dependence on dialysis (at least 3 sessions over at least 90 days); Diagnosis records of kidney failure or CKD stage 5; Record of kidney transplant
Incidence rate of a composite cardiovascular outcome in participants with CKD and T2D that initiate finerenone. | From first prescription/dispensation of finerenone (index date) until end of follow-up (death, disenrollment, development of either kidney failure or kidney cancer, or by the last available date in the corresponding database) up to 150 months
  Acute myocardial infarction, identified as an inpatient hospital diagnosis of fatal or non-fatal acute myocardial infarction. Congestive heart failure, identified as an impatient hospital or emergency department diagnosis of heart failure and stratified by new-onset or recurrent heart failure.
Drug utilization patterns in a cohort of participants with CKD and T2D that initiate finerenone. | From first prescription/dispensation of finerenone (index date) until end of follow-up (death, disenrollment, development of either kidney failure or kidney cancer, or by the last available date in the corresponding database) up to 150 months
  Depending on the database used, this includes incidence of drug use, initiation of treatment measured by drug prescription, drug dispensation, or a combination of both depending on data availability, dosing regimen, treatment persistence and non-persistence, and implementation measured as the proportion of days covered.
Number of participants who initiate finerenone at a 10 mg dose daily | At day 0 (first prescription/dispensation of finerenone)
Proportion of participants who continue the original 10 mg dose daily at the 1, 3, 6, and 12 months mark | From first prescription/dispensation of finerenone (index date) until 12 months after index date
Proportion of participants who up-titrate from 10 mg daily dose to a 20 mg dose daily at the 1, 3, 6, and 12 months mark | From first prescription/dispensation of finerenone (index date) until 12 months after index date
Number of participants who initiate finerenone at a 20 mg dose daily | At day 0 (first prescription/dispensation of finerenone)
Proportion of participants who continue the original 20 mg dose daily at the 1, 3, 6, and 12 months mark | From first prescription/dispensation of finerenone (index date) until 12 months after index date
Proportion of participants who down-titrate from 20 mg daily dose to a 10 mg dose daily at the 1, 3, 6, and 12 months mark | From first prescription/dispensation of finerenone (index date) until 12 months after index date
Incidence rate of hospitalization for heart failure in participants with CKD and T2D that initiate finerenone. | From first prescription/dispensation of finerenone (index date) until end of follow-up (death, disenrollment, development of either kidney failure or kidney cancer, or by the last available date in the corresponding database) up to 150 months
  Congestive heart failure, identified as an impatient hospital or emergency department diagnosis of heart failure and stratified by new-onset or recurrent heart failure.
Incidence rate of atrial fibrillation or flutter in participants with CKD and T2D that initiate finerenone. | From first prescription/dispensation of finerenone (index date) until end of follow-up (death, disenrollment, development of either kidney failure or kidney cancer, or by the last available date in the corresponding database) up to 150 months
Incidence rate of hyperkalemia in participants with CKD and T2D that initiate finerenone. | From first prescription/dispensation of finerenone (index date) until end of follow-up (death, disenrollment, development of either kidney failure or kidney cancer, or by the last available date in the corresponding database) up to 150 months
Incidence rate of hospitalization associated with hyperkalemia in participants with CKD and T2D that initiate finerenone. | From first prescription/dispensation of finerenone (index date) until end of follow-up (death, disenrollment, development of either kidney failure or kidney cancer, or by the last available date in the corresponding database) up to 150 months

CONTACTS AND LOCATIONS:
Locations (4):
- Many Locations, Multiple Locations, New Jersey, United States
- Bayer, Berlin, Germany
- Many Locations, Multiple Locations, Japan
- Many Locations, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.